CLINICAL TRIAL: NCT03213808
Title: ANALYSIS OF HEALTH DATA COLLECTED SYSTEMATICALLY BY THREE HOSPITALS FOR THE VALIDATION OF THE CHAPTER "ALLERGY AND HYPERSENSITIVITY" IN THE FUTURE VERSION 11 OF THE WORLD HEALTH ORGANIZATION (WHO) INTERNATIONAL CLASSIFICATION OF DISEASES (CIM)
Brief Title: VALIDATION OF THE CHAPTER "ALLERGIES AND HYPERSENSITIVITY" OF THE INTERNATIONAL DISEASE CLASSIFICATION (CIM)
Acronym: AHCIM11
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: UF9863
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-07

CONDITIONS: ALLERGIC OR HYPERSENSITIVITY
Keywords: Allergic diseases; hypersensitivity; International Classification of Diseases (ICD); World Health Organization (WHO)
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- respiratory allergies: respiratory allergies (asthma, rhinitis)
  Interventions: Other: No intervention: analysis of health data from patients with
- skin allergies: skin allergies (dermatitis, urticarial, angioedema)
  Interventions: Other: No intervention: analysis of health data from patients with
- anaphylaxis: anaphylaxis
  Interventions: Other: No intervention: analysis of health data from patients with
- gastrointestinal allergic conditions: gastrointestinal allergic conditions
  Interventions: Other: No intervention: analysis of health data from patients with
- ocular allergies: ocular allergies (conjunctivitis)
  Interventions: Other: No intervention: analysis of health data from patients with

INTERVENTIONS:
Other: No intervention: analysis of health data from patients with — No intervention: analysis of health data from patients with respiratory allergies (asthma, rhinitis), skin allergies (dermatitis, urticarial, angioedema), anaphylaxis, gastrointestinal allergic conditions and ocular allergies (conjunctivitis) for the validation of the chapter allergies and hypersensitivity in the future version of the WHO CIM

SUMMARY:
Allergic diseases, including allergic asthma, allergic rhinitis and anaphylaxis are not properly classified in current classifications of diseases. We here propose a project based on the evaluation of medical records of hospital databases of patients suffering for allergic and hypersensitivity conditions coded with the current and a new coming version of the international classification of diseases, no patient or intervention will be analysed.

We here propose a study to update and reach quality assurance of the classification of allergic and hypersensitivity conditions in international classification systems. The Allergic and hypersensitivity conditions section has indeed been recently built into the new ICD-11 framework and we aim to reach its quality assurance by evaluating medical records of French hospital databases. All the consecutive cases related to allergic and hypersensitivity conditions registered in the last 1 year will be selected and blind-coded by two independent coders based on the online English versions of the ICD-10 (2015 version) and ICD-11 Beta draft. The generated data will support the intra and inter-variability testing, survey among end-users and economic-impact evaluation. The economic impact of the transition from ICD-10 to ICD-11 will be analysed based on average estimated cost per day of each principal diagnosis and the effect of the classification change will be quantified by the cost variance of inter or intra diagnosis of ICD-10 and ICD-11. For the bridge procedure based on the alignment of the allergic and hypersensitivity conditions described into the ICD-10 (and ICD-10 CM US adaptation) framework to the ICD-11 beta phase, we propose the mapping and cross-linking terms methods. Meanwhile, we will start updating the allergic and hypersensitivity procedures by influencing the International Classification of Health Intervention (ICHI).

DETAILED DESCRIPTION:
Rationale for this Non-Interventional Study Allergic diseases, including allergic asthma, allergic rhinitis and anaphylaxis are not properly classified in current classifications of diseases. We here propose a project based on the evaluation of medical records of hospital databases of patients suffering for allergic and hypersensitivity conditions coded with the current and a new coming version of the international classification of diseases, no patient or intervention will be analized.

Objectives of this Non-Interventional Study Main Objectives: To assess the stability of codes for ICD-10 allergic diseases and hypersensitivity to ICD-11 using the medical-administrative databases of 3 hospitals.

Secondary Objectives: (I) To adjust the terms and links for allergic diseases and hypersensitivity and thus continue the on-line implementation process of ICD-11 based on the lessons learned on the main objective; (II) To estimate the economic impact of ICD-10 and ICD-11 transition for health care facilities; (III) To electronically align ICD-10 codes (and CM adaptation in the USA) with ICD-11.

Study design All the consecutive cases of allergies over a year and registered in the DIM bases of 3 healthcare establishments (the university hospital of Montpellier (CHRUM), Paris (APHP), Toulouse) will be individualized. Depending on the size of the facility, ½ to 1/10 of the cases will be included in the study. All cases will be selected anonymously. Two professional coders will encode the selected cases twice. The analysis of the data will be based on the degree of inter-encoder agreement using Cohen's Kappa coefficient. At the end of this process, we will be able to identify the correspondence between the codes recorded in the DIM database (ICD-10) and those of the new classification. In the event of discordant results, consensus will be reached by involving other coding experts from CHRUM. The economic impact of the transition from ICD-10 to ICD-11 will be approximated by estimating the average costs per ICD code used in the main diagnosis.

Target subject population Our project is focused on allergic and hypersensitivity sufferers. Although we intend to validate the classification of allergic and hypersensitivity conditions, the international classification systems are for global use and our methodology might be helpful for other diseases and for the program of medicalization and information system (PMSI).

Statistical methods In order to reach the inter and intra-variability testing, the data analysis will be based on the degree of inter-rater agreement using Cohen's Kappa.

The economic impact of the transition from ICD-10 to ICD-11 will be analized based on average estimated cost per day of each principal diagnosis and the effect of the classification change will be quantified by the cost variance of inter or intra diagnosis of ICD-10 and ICD-11.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

- We here propose a study based on hospital database medical records. The cases will be selected based on pre-established (ICD-10) allergy corresponding codes: respiratory allergies (asthma, rhinitis), skin allergies (dermatitis, urticarial, angioedema), anaphylaxis, gastrointestinal allergic conditions and ocular allergies (conjunctivitis).

The prescription of the medicinal product is clearly separated from the decision to include the subject in the non-interventional study

Exclusion criteria:

- We will exclude from the study all cases in which the ICD-10 codes are not related to allergic and hypersensitivity conditions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ALLERGIC OR HYPERSENSITIVITY CONDITIONS: respiratory allergies (asthma, rhinitis), skin allergies (dermatitis, urticarial, angioedema), anaphylaxis, gastrointestinal allergic conditions and ocular allergies (conjunctivitis)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Intra and inter-variability measures among coders and accuracy rate calculation | 1 day
  Ease of use, level of ambiguity on a 0-4 scale

SECONDARY OUTCOMES:
International Classification of Diseases -10, -10CM and -11 term alignement | 1 day
  International Classification of Diseases -10, -10CM and -11 term alignement

OTHER OUTCOMES:
Insertion of allergy procedures in the International Classification of Health Interventions (ICHI) | 1 day
  Insertion of allergy procedures in the International Classification of Health Interventions (ICHI)
Health economics related the transition from the ICD-10 to ICD-11: cost variance of inter or intra diagnosis of ICD-10 and ICD-11 | 1 day
  Health economics related the transition from the ICD-10 to ICD-11: cost variance of inter or intra diagnosis of ICD-10 and ICD-11

CONTACTS AND LOCATIONS:
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC